CLINICAL TRIAL: NCT05043675
Title: Director of Nuclear Medicine Department
Brief Title: Clinical Evaluation of [18F]APN-1607 PET Uptake in Alzheimer's Disease Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, FengWang, Director of nuclear medicine department, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: wf-[18F]APN-1607
Record Dates: First submitted 2021-09-13; First posted 2021-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]APN-1607 (Experimental): For the injection, subjects will receive a target dose of 0.1~0.15mCi/Kg [18F]APN-1607 as a bolus injection.
  Interventions: Drug: [18F]APN-1607

INTERVENTIONS:
Drug: [18F]APN-1607 — Subjects will receive one injection of [18F]APN-1607 (0.1~0.15mCi/Kg), a PET radiopharmaceutical selective for fibrillar tau. [18F]APN-1607 injection will be followed by a 10 ml saline flush.
  Other Names: [18F]PBB3

SUMMARY:
The overall objective of this study is to evaluate the overall pattern of [18F]APN-1607 uptake in subjects with AD dementia

DETAILED DESCRIPTION:
* To expand the safety and tolerability profile for the administration of [18F]APN-1607 and PET scanning.
* To assess regional patterns of [18F]APN-1607 uptake.
* To evaluate the relationship between regional measures of [18F]APN-1607 uptake and measurements of AD disease severity, such as National Institute on Aging and Alzheimer's Association (NIA-AA) diagnosis, Mini-mental Status Exam (MMSE) score, and Alzheimer's Disease Assessment Scale-cognitive subscale (ADAScog).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 45 to 80 years, inclusive.
* Has a diagnosis of AD dementia according to NIA-AA criteria, including significant impairment of activities of daily living.
* Has a CDR score ≥ 0.5 at screening.
* Has a MMSE score ≤ 25.
* Brain MRI supports the diagnosis of AD and there is no evidence of other nervous system diseases.
* Medications taken for symptomatic treatment of AD must have been stable for 30 days prior to screening and through completion of the neuropsychological battery.
* If necessary, the subject can be accompanied by nursing staff.
* Written informed consent must be obtained before any assessment is performed.
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year (ie, 12 consecutive months with no menses without an alternative medical cause) or, if they are of childbearing potential, must commit to use a barrier contraception method or to abstinence for the duration of the study and must have negative serum and urine pregnancy tests.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method (ie, condom), or to abstinence for the study duration.
* Male subjects must not donate sperm for the study duration.
* Willing and able to participate in all study procedures.

Exclusion Criteria:

* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Implants, such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.
* Intolerance to MRI noise or hermetic phobia.
* Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds local guidelines, eg, above an effective dose of 50 mSv.
* Current or prior history (within the last 10 years) of alcohol or drug abuse.
* Pregnant, lactating or breastfeeding.
* Unsuitable veins for repeated venipuncture
* Has received any investigational drug or device for any purpose within 30 days of screening (or 5 half-lives of the drug, whichever is longer).
* Known hypersensitivity to [18F]APN-1607 or its excipients
* Has received a non-vaccine investigational treatment for Aβ within the last 3 months.
* Has received a non-vaccine investigational treatment for tau within the last 3 months.
* Any situation that the presiding officer of this study believes may cause harm or potential harm to any link related to this test.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of [18F]APN-1607 Uptake Patterns by Regional SUV Values | 36 months
  [18F]APN-1607 uptake patterns will be assessed in regions of interest (ROIs) which relevant to AD pathology. Standard uptake value (SUV) will be calculated for each ROI, and standardized uptake value ratios (SUVRs) will be calculated by normalizing SUV of ROIs to the SUV of relevant reference region.

SECONDARY OUTCOMES:
Safety and Tolerability Profile Measured by Adverse Events (AEs) | 36 months
  Safety and tolerability profile for the administration of [18F]APN-1607 and positron emission tomography (PET) scanning are measured by number of participants with adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Study Director — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No